CLINICAL TRIAL: NCT00757250
Title: A Phase I Evaluation of the Safety and Biologic Activity of TXA127 in HIV-Infected Subjects With CD4+ T-Lymphocyte Counts Less Than 250 Per mm3 Who Have Responded to HAART
Brief Title: Safety Study of TXA127 to Elevate CD4+ T-Lymphocyte Counts in HIV-Infected Patients on Stable HAART Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty recruiting subjects to dosing cohort 5.
Sponsor: US Biotest, Inc. (Industry)
Collaborators: Tarix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXA127-2008-001
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Human Immunodeficiency Virus; CD4+ T-lymphocytes; treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — angiotensin I (1-7)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Dose Cohort 1: 50 mcg/kg/day of TXA127
  Interventions: Drug: Angiotensin 1-7
- 2 (Experimental): Drug Cohort 2: 100 mcg/kg/day TXA127
  Interventions: Drug: Angiotensin 1-7
- 3 (Experimental): Drug Cohort 3: 200 mcg/kg/day TXA127
  Interventions: Drug: Angiotensin 1-7
- 4 (Experimental): Drug Cohort 4: 300 mcg/kg/day TXA127
  Interventions: Drug: Angiotensin 1-7
- 5 (Experimental): Extended dosing cohort at 300mcg/kg TXA127 for 2 x 28-day treatment cycles, with an extended follow-up period to week 34.
  Interventions: Drug: Angiotensin 1-7

INTERVENTIONS:
Drug: Angiotensin 1-7 — Once daily subcutaneous injection of 50, 100, 200 or 300 mcg/kg/day
  Other Names: TXA127

SUMMARY:
The purpose of this study is to test the safety of an investigational medication, TXA127, and its ability to increase T-lymphocyte counts, specifically CD4+ T-lymphocytes, in persons infected with human immunodeficiency virus who are taking highly active anti-retroviral therapy.

DETAILED DESCRIPTION:
This is a Phase I, single institution, open-label, within-dosing-cohort-schedule randomized, dose escalation study of TXA127 in HIV-infected subjects with CD4+ T-lymphocyte counts less than 250 per mm3 who have responded to highly active retroviral therapy (HAART). The study has been designed to determine the maximum tolerated dose (MTD) of TXA127 in this subject population. This study will also obtain safety and biologic activity information about the subcutaneous injection of TXA127.

Five escalating dosing cohorts will be examined to determine the MTD. The first four dosing cohorts will receive 50, 100, 200 and 300 mcg/kg of TXA127 by subcutaneous injection daily for 14 days, followed by 14 days without treatment. These 28 days will be defined as one cycle. The cycle of therapy will be repeated once, for a total of two courses of treatment. The 5th dosing cohort will receive 300 mcg/kg of TXA127 by subcutaneous injection daily for 28 days, then 14 days without treatment followed by an additional 28 days of TXA127 administration. Dose escalation to the next cohort of subjects will be permitted to the next higher dosing level provided the following criteria have been met.

A standard Simon Phase I dose escalation trial has been proposed. The MTD will have been exceeded if the proportion of subjects that develops the same or similar study-drug-related, DLT in an assigned dosing schedule equals 2/2, 2/3, 2/4, 2/5, and 2/6 subjects. The MTD is defined as the largest dose that <2 of 6 subjects experiences a DLT. Dose-limiting toxicity is defined as a study-drug-related grade 3 or 4 adverse event (AE).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected males or non-pregnant, non-breast-feeding females who are >= 18 years of age;
* CD4+ T-lymphocyte count less than 250 per mm3;
* Successful response to HAART (defined as an HIV RNA viral load of <50 copies per mL) for a minimum of one year preceding study enrollment.

Exclusion Criteria:

* Opportunistic infection within the 6 months prior to study enrollment
* Active tuberculosis or other mycobacterial infection
* Uncontrolled high blood pressure or congestive heart failure class III or IV
* Systemic glucocorticoid or immunomodulator therapy within 30 days of study entry
* Prior history of Kaposi's sarcoma
* Prior history of lymphoma
* Active substance abuse within the last 30 days
* Uncontrolled psychiatric disorders, including depression
* Abnormal or inadequate liver or renal function
* Inadequate bone marrow function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
HIV-1 RNA viral load count | 18 weeks and 34 weeks (cohort 5)

SECONDARY OUTCOMES:
CD4+ T-lymphocyte count | 18 weeks and 34 weeks (cohort 5)

CONTACTS AND LOCATIONS:
Overall Officials: Gere S diZerega, MD, Study Director — US Biotest, Inc.; Robert A Larsen, MD, Principal Investigator — University of California, Keck School of Medicine
Locations (3):
- United States (3):
  - LAC+USC Medical Center, Rand Schrader Clini, Los Angeles, California
  - UCSD Division of Infectious Diseases, San Diego, California
  - Harbor - UCLA Medical Center, Torrance, California